CLINICAL TRIAL: NCT01162447
Title: Comparison of Bone Morphogenetic Protein-4 and -7 Levels (BMP-4 and 7) in the Serum, Ovarian Follicle Aspirates and Ovarian Organ Culture Supernatants Between Healthy Controls and Patients With Polycystic Ovarian Syndrome (PCOS).
Brief Title: Comparison of Bone Morphogenetic Protein-4 (BMP-4) and 7 Levels Between Control and Polycystic Ovarian Syndrome (PCOS) Patients.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Responsible Party: Ozgur Oktem, V.K.V. American Hospital Women's health center
Other Study IDs: MAR.YC.2008.0276
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-02

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: BMP- 4 and 7, polycystic ovarian syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Microphthalmia, Syndromic 6

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples, ovarian tissue samples, ovarian follicular fluid samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PCO: Healthy control subjects and patients with polycystic ovarian syndrome will be recruited for the study.

SUMMARY:
The investigators aim to compare the levels of bone morphogenetic protein-4 and -7 (BMP-4 and 7) in blood, follicular fluid and ovarian organ culture supernatant obtained from healthy subjects and polycystic ovarian syndrome (PCOS) patients.

DETAILED DESCRIPTION:
Female patients at ages 20-35 diagnosed with polycystic ovarian syndrome and age-matched healthy control subjects will be enrolled in this study.

Blood samples will be obtained at early follicular phase during doctor's visit from PCOS patients and control subjects.If the patient is amenorrheic at the time of visit, both random blood samples and another sample at early follicular phase after induction of withdrawal bleeding with progesterone.

Follicular fluids will be retrieved during oocyte pick-up procedure in patients undergoing assisted reproduction for PCOS and control IVF patients whose infertility is not PCO related.

Samples from ovaries will be collected at operation from PCOS patients and control subjects if they already undergo any gynecologic laparotomi operations.

Collected samples will be cultured for 7 days and BMP-4 and -7 levels will be measured in the culture fluid of the samples using ELISA method.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects and PCOS patients at ages 20-35 will be recruited for the study.

Exclusion Criteria:

* Those with any metabolic or endocrine problems other than PCOS will be excluded from the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who present to the women's health center of American Hospoital for complaints due to polcystic ovarian syndrome will be enrolled. Age-matched healthy subjects will be chosen for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Urman, MD, Study Director — VKV American Hospital Women's Health center
Locations (1):
- American Hospital Women's Health Center, Istanbul, Turkey (Türkiye)